CLINICAL TRIAL: NCT02951468
Title: Mid-term Outcome Following Revision Surgery of Clavicular Non- and Malunion Using Anatomic Locking Compression Plate and Iliac Crest Bone Graft
Brief Title: Mid-term Outcome Following Revision Surgery of Clavicular Non- and Malunion
Acronym: Nonunion
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Chlodwig Kirchhoff, PD Dr. med., Technical University of Munich
Other Study IDs: Beiromat_04
Record Dates: First submitted 2016-10-23; First posted 2016-11-01 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-10

CONDITIONS: Fracture, Healed, Fibrous Union
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nonunion group: All patients who were treated for clavicular non- or malunion with a locking compression plate and an iliac crest bone graft between January 2010 and December 2014 were included in this retrospective study.
  Interventions: Procedure: LCP plus iliac crest autograft

INTERVENTIONS:
Procedure: LCP plus iliac crest autograft — After exposure of the non- or malunion a complex multidimensional osteotomy of the clavicle with medial and lateral axial correction up to vital bone was performed [14]. Vital bone was verified by local blood extravasation resulting from drilling the previously osteotomized bone segments. The tricortical iliac crest bone graft was harvested according to the size assessed in the preoperative CT scan, consecutively adapted to the intraoperative measured size of the bony defect. After implantation of the bone graft the LCP was centered onto the clavicular shaft.

SUMMARY:
Background Treatment of clavicular non- and malunion is still challenging. Current surgical procedures often result in partially frustrating functional outcome along with high-grade subjective impairment and increased rates of revision surgery. However, the combination of vital bone graft and a biomechanically sufficient fixation system seems to be a promising concept of treatment.

Methods In this retrospective study, 14 patients with a mean age of 44 years (26-67 years) suffering from non-union (n=11) and/or malunion (n=4) of the clavicle were enrolled. All patients were surgically treated using an anatomical precontoured locking compression plate (LCP) and autologous iliac crest bone graft. Functional outcome was assessed using the age- and sex-specific relative Constant Score.

DETAILED DESCRIPTION:
Methods

Patients and follow-up

All patients who were treated for clavicular non- or malunion with a locking compression plate and an iliac crest bone graft between January 2010 and December 2014 were included in this retrospective study. The study protocol was approved by the local ethics committee (71/15 S).

The preoperative symptoms included pain (n=12), limited range of motion (n=2), pain when sleeping on the affected side (n=2), skin irritation caused by dislocated screws (n=1), feeling of weakness of the arm (n=1) and crepitation (n=1).

Standard radiographs of the affected clavicle (anterior-posterior path of rays perpendicular to radiographic cassette, anterior-posterior path of rays 30° tilted cephalad) were performed at the time of the initial presentation of the patient as well as during the routine follow-up examinations in our outpatient clinic. Preoperative planning included the performance of a magnetic resonance imaging (MRI) scan to estimate the non-vital parts of bone to be resected as well as the performance of a computed tomography (CT) scan of both clavicles to measure the original clavicle length to be able to adequately decide if a bone graft would be required. A tricortical iliac crest bone graft was used in all cases with bony defects larger than 15 mm due to the risk of abnormal shoulder biomechanics following clavicular shortening possibly resulting in pain, shoulder motion impairment and loss of strength.

The Constant Score was used to assess the shoulder function and activity preoperatively as well as during the routine follow-up examinations in our outpatient clinic. Subsequently the original Constant Score values were converted according to Gerber et al. to receive a normative age- and sex-specific Constant Score (relative Constant Score).

The implant

The LCP (locking compression plate) superior anterior clavicle plate with lateral extension (Depuy) is an anatomically precontoured fixation system with three to eight medial shaft holes for 3.5 mm locking or 3.5 mm cortex screws and six lateral 2.7 mm divergent locking or 2.4 mm cortex screws. This implant was used for treatment of all enrolled patients.

Surgical technique and rehabilitation

All patients underwent surgery placed in a beachchair position with the affected arm in a mobile position. A longitudinal skin incision was set below the clavicle with subsequent incision through the clavi-pectoral fascia also in longitudinal direction to allow for a later closure to ensure sufficient soft tissue coverage. After exposure of the non- or malunion a complex multidimensional osteotomy of the clavicle with medial and lateral axial correction up to vital bone was performed. Vital bone was verified by local blood extravasation resulting from drilling the previously osteotomized bone segments. The tricortical iliac crest bone graft was harvested according to the size assessed in the preoperative CT scan, consecutively adapted to the intraoperative measured size of the bony defect. After implantation of the bone graft the LCP was centered onto the clavicular shaft. At least three screws should be placed medially and laterally to the bone graft to ensure sufficient biomechanical stability. Before drilling the screw holes the plate position was controlled by fluoroscopy. If necessary the iliac crest bone graft should additionally be fixed by a suture cerclage (Fiber- Wire, Arthrex). After a final radiographical examination the wound was closed layer by layer.

Regarding postoperative rehabilitation primarily the affected arm was immobilized in a sling for 6 weeks. Patients started physiotherapy on the first postoperative day following a standard rehabilitation protocol: abduction and flexion were restricted to 30° for the first two weeks, to 60° for the week three and four postoperative and to 90° for week five and six postoperative. Full weight bearing was not allowed before week 12 postoperative. 3, 6, 12 and 24 weeks postoperatively radiographs were performed to evaluate bone healing.

ELIGIBILITY:
Inclusion Criteria:

* clavicular non-unions or malunions

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from clavicular non-unions or malunions
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change of Functional Outcome in comparison to preoperative state | 1,5 yrs.
  Shoulder Function, assessed by MSQ

IPD SHARING:
Plan to Share IPD: No
No Plan